CLINICAL TRIAL: NCT02166086
Title: Advanced Imaging for Diagnosing Pancreatico-biliary Disorders: A Multicenter Registry.
Brief Title: Advanced Imaging Registry for Diagnosing Pancreatico-biliary Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief of Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1111012020
Record Dates: First submitted 2014-06-10; First posted 2014-06-18 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diagnosis of a Pancreaticobiliary Disorder
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic imaging: Any patient who has undergone advanced imaging procedures for diagnosis and/or treatment of a pancreatico-biliary disorder.
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Endoscopy involving advanced imaging techniques

SUMMARY:
The purpose of this registry is to record information and evaluate the impact of advanced imaging techniques on the management of pancreatico-biliary disorders. The registry will evaluate diagnostic performance and overall clinical management impacted by advanced imaging techniques.

DETAILED DESCRIPTION:
Advanced imaging techniques such as SpyGlass or pCLE (probe-based Confocal laser endomicroscopy) using Cellvizio probes enable high sensitive and specific diagnosis of strictures or tumors in bile and pancreatic ducts. However, advanced endoscopists have only recently started to employ such techniques for diagnostic purposes. Hence we lack enough data to evaluate the sensitivity, specificity, accuracy, technical feasibility and safety of such imaging devices. Evaluation of these factors would help us compare them to conventional diagnostic options; and consequently help us identify appropriate advanced imaging techniques for biliary and pancreatic disorders and improve clinical management of patients.

The purpose of this registry is to record information and evaluate the impact of advanced imaging techniques on the management of pancreatico-biliary disorders. The registry will evaluate diagnostic performance and overall clinical management impacted by advanced imaging techniques.

This multi-center registry has been initiated:

* To document the impact of advanced imaging techniques in pancreatico-biliary disorders on the clinical management of pancreatico-biliary disorders including malignancies.
* To assess the sensitivity, specificity, accuracy, technical feasibility and safety of advanced imaging techniques in pancreatico-biliary disorders.

The registry will review and document:

* All patients who have had advanced imaging done for pancreatico-biliary disorders.
* No subject intervention is involved in this study. Subject contact is not needed for database review.

Study Design at Secondary sites:

* Other sites must have either a database review protocol and/or a clinical trial that would collect data on advanced imaging done for pancreatico-biliary disorders prior to participating in the registry.
* These sites would have IRB approved protocols to collect and send advanced imaging procedure data to the primary site (WCMC). Additionally, the secondary study sites would mention WCMC as an entity that could receive PHI in their respective protocols and consent/HIPAA forms.
* All secondary study sites' IRB approvals will be sent to the primary/coordinating study center at WCMC. The primary center will then forward these IRB approvals to WCMC IRB as soon as they are received from the secondary study sites.
* Relevant IRB documentation will be maintained at both primary and secondary sites.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has undergone advanced imaging procedures for diagnosis and/or treatment of a pancreatico-biliary disorder.
* Above 18 years of age.

Exclusion Criteria:

* Any patient who has not undergone advanced imaging techniques for pancreatico-biliary disorders.
* Below 18 years of age.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who has undergone advanced imaging procedures for diagnosis and/or treatment of a pancreatico-biliary disorder.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-09; Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy Profile | 1 year
  Documentation of accuracy, sensitivity, specificity, positive predictive value, negative predictive value based on final diagnosis variable analyses.

SECONDARY OUTCOMES:
Survival duration | 1 year or more
  Documentation of follow up diagnoses variable and survival duration (in days).

OTHER OUTCOMES:
Efficacy | 1 year
  Documentation of technical success and clinical success rates. Technical success will be recorded as procedure success and capturing of relevant advanced imaging. Clinical success will be recorded as if a diagnosis was made based on the advanced imaging results.
Safety Profile | 30 days
  Documentation of Safety: Number of Participants with Adverse Events; Type, frequency and intensity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD sharing

REFERENCES:
- [Derived] Tyberg A, Xu MM, Gaidhane M, Kahaleh M. Second generation optical coherence tomography: Preliminary experience in pancreatic and biliary strictures. Dig Liver Dis. 2018 Nov;50(11):1214-1217. doi: 10.1016/j.dld.2018.05.019. Epub 2018 Jun 8. PMID 29937365
- [Derived] Karia K, Waxman I, Konda VJ, Gress FG, Sethi A, Siddiqui UD, Sharaiha RZ, Kedia P, Jamal-Kabani A, Gaidhane M, Kahaleh M. Needle-based confocal endomicroscopy for pancreatic cysts: the current agreement in interpretation. Gastrointest Endosc. 2016 May;83(5):924-7. doi: 10.1016/j.gie.2015.08.080. Epub 2015 Sep 14. PMID 26382051
- [Derived] Karia K, Jamal-Kabani A, Gaidhane M, Tyberg A, Sharaiha RZ, Kahaleh M. Probe-Based Confocal Endomicroscopy in Primary Sclerosing Cholangitis: Not All Inflammatory Strictures Are the Same. Dig Dis Sci. 2016 Jan;61(1):283-6. doi: 10.1007/s10620-015-3827-1. Epub 2015 Aug 2. PMID 26233552